CLINICAL TRIAL: NCT02397863
Title: An Open Label, Multi-Center Study to Investigate the Safety of Cannabinoid (GWP42003-P) in Children With Medication Resistant Epilepsy
Brief Title: Epidiolex and Drug Resistant Epilepsy in Children
Acronym: CBD
Status: Available | Type: Expanded Access
Sponsor: Augusta University (Other)
Collaborators: State of Georgia (Unknown)
Responsible Party: Principal Investigator, Yong Park, Professor Child Neurology, Professor Pediatrics, Augusta University
Other Study IDs: CBD02
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol (Epidiolex) — Daily dosage up to 25 mg/kg/day with an optional up titration to a maximal daily dosage up to 50 m/kg/day until End of Treatment.
  Other Names: Epidiolex

SUMMARY:
This open-label, multi-center study is open to patients 1 to 18 years of age at time of enrollment with medication resistant epilepsy.

DETAILED DESCRIPTION:
This open-label, multi-center study is open to patients 1 to 18 years of age at time of enrollment with medication resistant epilepsy. The study consists of an 8 week baseline, titration, and treatment of Epidiolex in a daily dosage up to 25 mg/kg/day, with an optional secondary titration schedule after 26 weeks of treatment up to a maximal daily dosage up to 50 m/kg/day until End of Treatment, followed by a taper-down period, and a safety follow up. Treatment will be provided for a total of 52 weeks with an interim analysis conducted 12 weeks after achieving maximal dose (either 25 mg/kg/day or optimal dose with regards to safety and tolerability) and at the end of 1 year of treatment with treatment extensions conducted beyond 52 weeks until such time as there is market authorization for Epidiolex, if Epidiolex becomes unavailable, or the study is terminated. Cessation of Epidiolex administration will be concluded with a taper period and follow-up visit 4 weeks after the taper.

ELIGIBILITY:
Inclusion Criteria:

* Patient should have history of trying at least four antiepileptic drugs (AEDs), including one trial of a combination of two concomitant drugs, without successful seizure control. Vagal nerve stimulation, RNS deep brain stimulation, or the ketogenic diet can be considered equivalent to a drug trial.
* Patient must be taking two or more AEDs at a dose which has been stable for at least four weeks.
* A State of Georgia resident.

Exclusion Criteria:

* Patient is diagnosed as having Dravet Syndrome or Lennox-Gastaut Syndrome and eligible for a GW Pharmaceutical-Sponsored Clinical Trial.
* Patients who have been part of a clinical trial involving another investigational product in the previous six months.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2014-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yong D Park, MD, Principal Investigator — Professor
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States